CLINICAL TRIAL: NCT01067534
Title: Assessment of Bronchodilator Responsiveness in Healthy Young Adults Using Forced Oscillations
Brief Title: Bronchodilator Responsiveness in Healthy Young Adults Using Forced Oscillations Technique (FOT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Patras (Other)
Responsible Party: Michael Anthracopoulos, Assoc. Prof. of Pediatrics and Pediatric Pulmonology, University of Patras, Patras, Greece
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: FOT_PATR_2010
Record Dates: First submitted 2010-02-10; First posted 2010-02-11 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2010-04

CONDITIONS: Bronchodilation
MeSH Terms: interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Salbutamol — Inhaler salbutamol 0,1 mg/dose - 4 doses=0,4 mg
  Other Names: Aerolin

SUMMARY:
Studies evaluating response to bronchodilation in flow-volume spirometry and/or by forced oscillations technique (FOT), have been conduced in subjects with obstructive airways diseases. Less is known about bronchodilation responses, assessed by both spirometry and FOT in healthy young subjects.

The purpose of the present study is

1. to determine the range of the bronchodilation response in terms of changes in selected spirometric parameters in healthy non-smoking young adults, for identifying normal response after an inhaled bronchodilatory agent versus placebo, and its anthropometric and spirometric determinants
2. to determine the range and characteristics of bronchodilation response using pseudorandom FOT in healthy non-smoking young adults, for identifying normal response after an inhaled bronchodilatory agent versus placebo, and its anthropometric and oscillometric determinants.
3. to compare and correlate eventual changes in spirometric and oscillometric parameters.

The investigators hypothesize that exists a normal variation in spirometric and oscillometric parameters after bronchodilation, and that these parameters are correlated.

DETAILED DESCRIPTION:
INTRODUCTION

Studies evaluating response to bronchodilation in flow-volume spirometry and/or by forced oscillations technique (FOT), have been conduced in subjects (children or adults) with obstructive airways diseases. Less is known about bronchodilation responses, assessed by both spirometry and FOT in healthy young subjects.

PURPOSE

The purpose of the present study is

1. to determine the range of the bronchodilation response in terms of changes in PEF, FEV1, FEF25, FEF50, FEF75, and FEF25-75, in healthy non-smoking young adults, for identifying normal response after an inhaled bronchodilatory agent versus placebo, and its anthropometric and spirometric determinants
2. to determine the range and characteristics of bronchodilation response using pseudorandom FOT in healthy non-smoking young adults, for identifying normal response after an inhaled bronchodilatory agent versus placebo, and its anthropometric and oscillometric determinants.
3. to compare and correlate eventual changes in spirometric and oscillometric parameters.

MATERIAL AND METHODS

The study will be conduced in the Laboratory of Respiratory Functions of the University Hospital of Patras, Patras, Greece.

Healthy, non-smoking young adults (medical students and residents) will be voluntary included. Participants will be assessed for eligibility with a structured interview which include questions regarding respiratory symptoms (wheezing, attacks off shortness of breath, sputum production, and dyspnea at rest or on exertion), diagnosed respiratory diseases, and use of pulmonary medication. A subject will be considered as non-smoker if he/she has never smoked or has discontinued smoking at least 5 years prior to entering the study.

Anthropometric data will be obtained at the enrollment. All oscillometric and spirometric measurements will be performed during morning hours (09:00 to 12:00). Subjects will be advised to refrain from consuming coffee or tea, and engaging in heavy eating for 2 hours.

Respiratory impedance spectra (Zrs), yielding resistance (Rrs) and reactance (Xrs) as a function of frequency, will be obtained using a commercially available device (i2m, Chess Medical, Belgium), in accordance with the ERS 2003 guidelines. The forced oscillatory signal is a pseudorandom signal consisting of frequency components between 4 and 48 Hz with a measurement period of 8 sec. During measurement the subject will be seated comfortably upright with the neck in the neutral position and the arms resting comfortably by the side. The cheeks and lower jaw of the subject will be firmly supported by a staff member during all measurements. Participants will be connected to the device via a mouthpiece incorporating a bacterial filter and instructed to breathe normally with a nose clip in place. Five technically acceptable measurements will be obtained. A measurement will be considered unacceptable if coherence will be <0.95 at 2 or more frequencies or if Zrs show obvious artifacts. The calibration of the device will be checked daily with a known resistance. All measurements will be performed by the same trained respiratory physician.

Spirometric measurements will always follow FOT measurements. Spirometry will be completed with a flow-volume device (MasterScreen IOS, Viasys/Jaeger; Höchberg, Germany), with the subject seated, using ATS 1994 criteria for performing the maneuver. Nose clips and disposable bacterial filters will be used. At least three technically acceptable measurements will be recorded with a maximum of eight efforts. All measurements will be performed by the same trained respiratory physician. The calibration of the device will be checked daily with a 3-L calibration syringe (Viasys/Jaeger; Höchberg, Germany).

The subjects will inhale 0.4mg of salbutamol (Aerolin, GlaxoSmithCline, London, UK) through a spacer device (Volumatic, GlaxoSmithCline), or a placebo inhaler (Allen & Hanburys LTD, Greenford, UK) again through a similar spacer. Special measures will be taken to ensure the blindness of the participants regarding the received inhaler.

Respiratory function measurements (FOT followed by spirometry) will be repeated (as described above) 15 min after the inhalation. Subjects will remain seated without consuming beverages other than water.

Each subject will have two sessions of baseline and post-inhalation measurements; one after receiving salbutamol and one after placebo. These sessions will be performed one day apart. The respiratory physician who will perform the measurements will be unaware regarding the received inhaler.

All technically acceptable Zrs measurements will be averaged and mean Rrs and Xrs at 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30, 32, 34, 36, 38, 40, 42, 44, 46, and 48 Hz will be calculated. The resonance frequency, the average Rrs between 4-24 Hz (Rrs 4-24) and 4-48 Hz (Rrs 4-48), and the frequency dependence of Rrs 4-24 and Rrs 4-48 will be also assessed. Absolute and relative changes after bronchodilation or placebo will be examined.

Spirometric variables which will used in analysis will include PEF, FEV1, FEF25, FEF50, FEF75, and FEF25-75. Absolute and relative changes after bronchodilation or placebo will be examined.

Multiple linear regression analysis will be performed to determine the individual effects of the following factors on absolute and relative bronchodilatory responses: age, sex, height, weight, BMI, and baseline lung function. The Pearson correlation will be used to assess the association of oscillometric and spirometric variables. All analyses will be performed using SPSS 17 for windows (SPSS, Chicago, IL).

ELIGIBILITY:
Inclusion Criteria:

* Healthy non-smoking young adults

Exclusion Criteria:

* Respiratory symptoms
* Respiratory disease
* Respiratory medication
* Smoking

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Bronchodilation responses, assessed by both spirometry and FOT, in healthy young subjects after receiving salbutamol or placebo | 15 minutes after inhalation of salbutamol or placebo

CONTACTS AND LOCATIONS:
Overall Officials: Michael Anthracopoulos, MD, Study Director — University Hospital of Patras, Greece; Sotirios Fouzas, MD, Principal Investigator — University Hospital of Patras, Greece; Konstantinos Bolis, MD, Principal Investigator — University Hospital of Patras, Greece
Locations (1):
- University Hospital of Patras, Pátrai, Greece